CLINICAL TRIAL: NCT06330142
Title: T-QAP: radioTherapy eQuicie Adolescent - Pediatrics
Brief Title: Hippotherapy Teenager-pediatric Radiotherapy
Acronym: T-QAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Paul Strauss (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-006
Record Dates: First submitted 2024-03-07; First posted 2024-03-26 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Radiotherapy
Keywords: Radiotherapy; Equicie; Adolescent; Pediatric

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- entire study population (Other)
  Interventions: Other: Participation in 10 horse-assisted therapy sessions

INTERVENTIONS:
Other: Participation in 10 horse-assisted therapy sessions — supporting children and teenagers undergoing radiotherapy with a horse-assisted therapy approach

SUMMARY:
This study proposes a horse-assisted therapy (HAT) approach to accompany children and young adults undergoing irradiation in the ICANS Radiotherapy Department.

The aim of this new approach is to improve quality of life and reduce anxiety in children and adolescents treated with radiotherapy. The impact of equine-assisted therapy on quality of life and anxiety disorders will be described prospectively between the start and end of irradiation in children and parents who agree to inclusion.

DETAILED DESCRIPTION:
Electro-radiology medical technician (ERMT) are privileged contacts with children. They accompany them every day during radiotherapy sessions. An animal-mediated approach would provide a new out-of-hospital environment. The equine sessions, precious moments when the child can forget about his illness, would enable him to escape from his condition as a patient. Indeed, the sick child adopts a posture to withstand treatment and take on responsibilities such as "not crying" and "being brave". These moments, away from the hospital, are essential to the smooth running of care, since they limit the weariness induced by daily radiotherapy sessions and help preserve the quality of caregiver/child cooperation during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 to <18 years.
* With an indication for radiotherapy for cancer (of any type)
* Patients hospitalized and/or managed on an ambulatory basis
* WHO ≤ 2
* Child and parents (or accompanying adults) who speak and understand French
* Free, express and informed consent of the adult patient OR of those exercising parental authority for minor patients
* Child with social security coverage

Exclusion Criteria:

* Children afraid of horses and stables
* Contraindication to the practice of equine-assisted therapy (allergy to horses or dust, children with asthma attacks triggered by dust/animal hair ...)
* Patient on stretcher
* Children or parents (or carers) with significant cognitive impairment, making self-assessment or hetero-assessment impossible even with assistance
* Unavailability or lack of interest in participating in equine-assisted therapy sessions

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2027-06-19 (Estimated); Study Completion 2027-06-19 (Estimated)

PRIMARY OUTCOMES:
Evolution of quality of life between the beginning and the end of horse-assisted therapy (HAT) in children (self-questionnaire) treated with radiotherapy | before radiotherapy, halfway through the HAT sessions (at 5 weeks), at the end of the HAT sessions (at 10 weeks) and one month after the end of the HAT sessions
  The questionnaire used to assess quality of life will be completed by the child.
  Two versions of the VSP-A questionnaire exist, depending on the child's age (versions < 10 years and 10-17 years).
  Results can be compared with reference values for the general population.

SECONDARY OUTCOMES:
Improving children's quality of life between the start and end of irradiation (hetero-questionnaire) by HAT | before radiotherapy, halfway through the HAT sessions (at 5 weeks), at the end of the HAT sessions (at 10 weeks) and one month after the end of the HAT sessions
  Parents (or carers) will complete a questionnaire to assess their child's quality of life.
Decrease anxiety disorders between the beginning - child version and end of irradiation in children (self-questionnaire) with HAT | before radiotherapy, halfway through HAT sessions (at 5 weeks), at the end of HAT sessions (at 10 weeks) and one month after the end of HAT sessions
  The questionnaire used to assess anxiety will be completed by the child (SCARED child version)
Decrease anxiety disorders between the beginning - parents' version and end of irradiation in children (self-questionnaire) with HAT | before radiotherapy, halfway through HAT sessions (at 5 weeks), at the end of HAT sessions (at 10 weeks) and one month after the end of HAT sessions
  Parents (or carers) will also complete a questionnaire to assess their child's anxiety (SCARED parents' version)
Assessing the acute side effects of radiotherapy at the start and end of irradiation | at the start and end of radiotherapy sessions (from 3 to 7 weeks)
  Evaluation of acute toxicities induced by radiotherapy CTCAE version 5 scale
Study the relevance of the various equestrian activities proposed as a strategy for improving care through the horse | At every HAT sessions (up to 10 weeks)
  Study the link between the various equestrian activities and the quality of life reported by children. Dashboard to track the duration of each activity carried out per child and per session, completed by the equestrian.
Evaluate participant's expectations and satisfaction with their care | at the beginning and end of HAT sessions (up to 10 weeks)
  questionnaire
Assess the medical electroradiology technician's (MERT's) impression of the child's well-being during irradiation | every week during radiotherapy (from 3 to 7 weeks)
  MERT's assessment of the impact of HAT on the child's well-being, based on a retrospective questionnaire for the previous week.
Assessing the impact of HAT on the child during irradiation according to the MERT | at each radiotherapy session (from 3 to 7 weeks)
Evaluate the rider's impression of the child's well-being of the child during HAT sessions | at the end of the first session and at the end of the last session of HAT (up to 10 weeks)
  Equestrian appreciation of the impact of HAT on the child's well-being during HAT sessions using questionnaires
Assessing the impact of an alternative activity on parents' satisfaction with care | at the end of the HAT sessions (at 10 weeks)
  Open questionnaire at the end of HAT to be completed by parents

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Paul Strauss, Strasbourg, France